CLINICAL TRIAL: NCT03038698
Title: Paediatric and Adult African Spirometry II: A Determination of Reference Equation in South African Children and Adults
Brief Title: Paediatric and Adult African Spirometry II
Acronym: PAASII
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of KwaZulu (Other)
Collaborators: AstraZeneca (Industry); Medical Research Council, South Africa (Other)
Responsible Party: Sponsor
Other Study IDs: BE295/16
Record Dates: First submitted 2017-01-30; First posted 2017-02-01 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-01

CONDITIONS: Lung Diseases
Keywords: spirometry; normative values; health; south africa; children
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Pulmonary function testing is the most widely used tool for the diagnosis, severity assessment, management, risk factor categorization and follow-up of individuals with chronic lung disease. Africa has a high burden of infectious respiratory diseases which include tuberculosis, asthma and human immunodeficiency virus-related lung disease. Coupled with this is an increasing burden of non-communicable respiratory diseases; which include chronic obstructive pulmonary disease, emphysema, bronchiectasis and asthma. A proviso to the use of lung function testing is the determination of "normal" values; which are determined for age, gender, height and ethnicity for the relevant population. It is well recognised that the comparison of an individual patients' results to an ethnically inappropriate population may lead to the under or -over diagnosis of disease, inappropriate treatments and result in increased burden on individuals, their families and the healthcare system.

The investigators therefore propose to conduct a prospective well-designed study to include a representative sample of both adults and children (4000); to verify the validity of the retrospective pilot data, in a South African population.

DETAILED DESCRIPTION:
Pulmonary function testing is the most widely used tool for the diagnosis, severity assessment, management, risk factor categorization and follow-up of individuals with chronic lung disease. Africa has a high burden of infectious respiratory diseases which include tuberculosis and human immunodeficiency virus-related lung disease.Coupled with this is an increasing burden of non-communicable respiratory diseases; which include chronic obstructive pulmonary disease, emphysema, bronchiectasis and asthma [1,2]. The management of these colliding epidemics requires correct diagnosis and management in order to ensure adequate resource allocation and avoidance of unnecessary costs.

A proviso to the use of lung function testing is the determination of "normal" values; which are determined for age, gender, height and ethnicity for the relevant population [3]. These "normal' values should also take into account the normal lung function decline associated and the aging process. It is well recognised that the comparison of an individual patients' results to an ethnically inappropriate population may lead to the under or -over diagnosis of disease, inappropriate treatments and result in increased burden on individuals, their families and the healthcare system [4-6]. There are numerous published reference equations, but the recently published Global Lung Initiative multi-ethnic reference equations published in 2012(GLI2012) collated the largest spirometry data set from individuals aged 2.5 to 95 years [7]. The innovation in GLI2012 was that it allowed for the smooth transitioning of data from childhood adulthood using sophisticated statistical modelling.

The investigators have previously collated data in phase 1 of this study using the GLI methodology on published African spirometry data from 26 594 individuals, and found a wide variation in predicted z-scores when fitting the African data to GLI2012, with a fairly good match between the black African males and African-Americans [15]. This dataset was skewed as due to the large number of African males and with a disproportionally larger contribution of data from North Africa and therefore requires confirmation. The investigators therefore propose to conduct a prospective well-designed study to include a representative sample of both adults and children (4000); to verify the validity of the retrospective pilot data, in a South African population.

ELIGIBILITY:
Inclusion Criteria:

* Study involves African adults and children age 5 to 95 years.
* Study number of at least 300 'healthy' subjects [7] per population band as per table 1.
* Availability of essential background information for each subject (birth date, date of test, gender, height, weight, body mass index, socioeconomic status and ethnic group).
* Consent given for adults 18 years and above, and assent for children over the age of 8 years and parental/guardian consent for all children under the age of 18 years.

Exclusion Criteria:

* Inter-current upper or lower respiratory tract infection
* Chronic lung diseases: including asthma and chronic obstructive pulmonary disease
* Current or previous tuberculosis infection
* Myocardial infarction
* Stroke
* Muscular disorders
* Previous history of cardiac diseases
* Current smoker
* Past smoker with >5 pack year of tobacco
* Previous lung surgery

Ages: 5 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study will be conducted in four regions in South Africa: KwaZulu Natal, Western Cape, Limpopo and Gauteng Province. Two sampling frames will be used with a paediatric and adult population. The paediatric sample frame will be school-going children (6 to 18 years) at primary and secondary schools during school days. For the adult sample, data will be collected on healthy adults age of 18 to 95 years, lung function testing will be conducted in conjunction with the South African Statistical Services (General Health Survey) a household surveys to ensure random population sampling from the four identified provinces from January 2016 to October 2017.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-12-30 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
lung function in healthy adults and children | 2 years
  lung function reference equations determination in healthy adults and children

CONTACTS AND LOCATIONS:
Locations (1):
- University of KwaZulu Natal, Durban, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: No
All results of the study will be published in a peer-reviewed journal